CLINICAL TRIAL: NCT01889888
Title: Effectiveness and Safety of Endoscopically-Assisted Submucosal Administration of Autologous Adipose-Derived Regenerative Cells for the Treatment of Urethral Strictures
Brief Title: Effectiveness and Safety of Autologous Adipose-Derived Regenerative Cells for the Treatment of Urethral Strictures
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Burnasyan Federal Medical Biophysical Center (Other Government)
Responsible Party: Principal Investigator, Pavel Kyzlasov, MD, Burnasyan Federal Medical Biophysical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-FMBC-01-02-13
Record Dates: First submitted 2013-06-25; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Urethral Strictures in Males
Keywords: Male urethral stricture; ADRC; Adipose-derived regenerative cells; Fat tissue; Stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADRC injection (Experimental)
  Interventions: Other: Submucosal injection of ADRC

INTERVENTIONS:
Other: Submucosal injection of ADRC — Subjects will undergo liposuction under local anesthesia. Lipoaspirate will be processed to isolate and concentrate ADRCs. Patients will undergo mechanical dilation followed by submucosal periurethral ADRC injections circle-wise into stricture site under endoscopic vision.

SUMMARY:
Autologous adipose-derived regenerative cells (ADRC) extracted using Celution 800/CRS System (Cytori Therapeutics Inc)from a portion of the fat harvested from the patient's front abdominal wall. ADRC will be administered one-time endoscopically into submucosal layer of urethra under eye control into the stricture site after mechanical dilation. This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Fat tissue obtainment. Subjects will undergo liposuction under local anesthesia. In this procedure, Ringer's solution with the anesthetic lidocaine and vasoconstrictor adrenaline infused into the adipose compartment to minimize blood loss and contamination of the tissue by peripheral blood cells. 15 minutes later a hollow blunt-tipped 3 mm cannula introduced into the subcutaneous space through small (0.5 cm) incision. The cannula attached to syringe and under gentle suction moved through the adipose compartment, mechanically disrupting the fat tissue. Aspirate volume - approximately 150-200 cc. Procedure time - 30 minutes.

ADRC isolation. Aspirated fat tissue placed into sterile vessel which inserted into Celution 800/CRS System (Cytori Therapeutics Inc) - closed system for automated and standardized extraction and concentration of ADRC. Celution 800/CRS System drains excess of fluid from fat tissue and estimate it's volume After that lipoaspirate washed extensively with equal volumes of Ringer's solution to remove blood. At the end of this process System indicates required volume of enzyme reagent (Celase®) which should be added immediately by operator. After enzyme treatment Celution 800/CRS System automatically transfers isolated ADRC into washing compartment where ADRC washed and concentrated in 5 mL suspension. Tissue processing time - approximately 60 minutes. ADRC suspension match all requirements listed in technical documentation for Celution 800/CRS System. Obtained ADRC divided into 2 portions. First portion (0.2-0.5 mL) used for counting, viability and sterility assessment. Second portion placed into sterile syringe for injection.

Urethral stricture dilation. Under direct vision HiWire® hydrophilic nitinol wire positioned through the urethra and exchanged for a stiff-bodied wire. After that S-Curve urethral dilators (Cook Medical Inc.) passed over the wire guide progressing from the smallest to the largest 24(Fr) appropriate size while maintaining the wire guide's position.

Periurethral injection of ADRC. After dilation needle for injection introduced into urethra using endoscope. Urethra punctured several times circle-wise at the region of stricture at depth of 5 mm under endoscopic vision and 0.3-0.5 mL of ADRC suspension injected submucosally each time. Total volume of solution injected depends on stricture length and technical possibilities. Minimal injected volume - 3 mL, maximal - 4.5 ml. After fat micrograft injected, urethral balloon catheter placed and removed the following day.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from urethral strictures at least for 1 year
* Moderate and severe grade of obstructive voiding symptoms according to assessment made by investigator
* Patient is familiar with Participant information sheet.
* Patient signed informed consent form

Exclusion Criteria:

-Contraindications for local anesthesia

For the patients undergone surgical treatment of prostate cancer:

* Cancer relapse
* prostate-specific antigen (PSA) level >0.008 ng/mL

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-10 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint-1 | 4 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse events (SAEs)
Safety endpoint-2 | 4 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse reactions (SARs)

SECONDARY OUTCOMES:
Efficacy endpoint-1 | 10 days, 4, 12, 24, 48 weeks after treatment
  Retrograde urethrogram
Efficacy endpoint-2 | 10 days, 4, 12, 24, 48 weeks after treatment
  Urodynamic studies: postvoid residual (PVR) volume measurement, uroflowmetry.
Efficacy endpoint-3 | 10 days, 4, 12, 24, 48 weeks after treatment
  Quality of life measured by the International Prostatic Symptom Score (IPSS) and the Short Form (36) Health Survey (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Ilya I Eremin, MD, PhD, Principal Investigator — Burnasyan Federal Medical Biophysical Center; Pavel S Kyzlasov, MD, Principal Investigator — Burnasyan Federal Medical Biophysical Center
Locations (1):
- State Research Center Burnasyan Federal Medical Biophysical Center FMBA of Russia; Center for Biomedical Technologies, Moscow, Russia